CLINICAL TRIAL: NCT07073378
Title: BCI@Home: Brain Computer Interface Solutions to Enable Youth Living With Severe Disabilities
Acronym: BCI@home
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Adam Kirton, Pediatric Neurologist, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB25-0495
Record Dates: First submitted 2025-06-24; First posted 2025-07-18 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy; Pediatric Stroke; Genetic Condition; Acquired Brain Injury (Including Stroke)
Keywords: pediatric brain computer interface
MeSH Terms: conditions — Cerebral Palsy; Genetic Diseases, Inborn; Brain Injuries | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCI at home (Experimental): Home BCI use. Families will first complete an in-person visit to review available activities, set their first goals, and learn to use BCI independently. A BCI "kit" will be given to each family, with a headset and the equipment and software required to pursue their identified goals. Following this, families will participate in 12 virtual sessions over 3-6 months. Scheduling will be flexible to accommodate complex family needs. Daily online support will be provided via a messaging application. Participants who choose to continue using BCI beyond 12 sessions will be provided kits and supported.
  Interventions: Device: Brain computer interface

INTERVENTIONS:
Device: Brain computer interface — Families will first complete an in-person visit to review available activities, set their first goals, and learn to use BCI independently. A BCI "kit" will be given to each family, with a headset and the equipment and software required to pursue their identified goals. Following this, families will participate in 12 virtual sessions over 3-6 months. Scheduling will be flexible to accommodate complex family needs. Daily online support will be provided via a messaging application. Participants who choose to continue using BCI beyond 12 sessions will be provided kits and supported.

SUMMARY:
The goal of this trial is to evaluate use of brain computer interfaces (BCI) at home for children with severe severe physical disabilities. The main questions it aims to answer are:

1. Can a home BCI program enable children with disabilities to achieve personalized life participation goals?
2. Can a home BCI program promote implementation reach?

DETAILED DESCRIPTION:
Preliminary research has proven that children with severe physical disabilities can operate home BCI systems. Despite the incredible impact of BCI on child well-being, access is currently limited to those who are close to major centres with the resources to frequently access tertiary care sites. A home-based BCI program is necessary to make this technology equitably available so that every child can realize their fundamental human right to participate in life.

The objectives are to: (1) Evaluate the effectiveness of a home BCI program for enabling children with disabilities to achieve personalized life participation goals; (2) Evaluate the equitable reach of implementation of a home BCI program.

This is a prospective, family-centered, single arm hybrid effectiveness-implementation trial that uses mixed methods. Implementation and effectiveness outcomes will be examined in parallel to ensure the program remains effective as its reach expands.

Implementation Methods: The trial uses systematic implementation science methods focused on the sustainable uptake of research into real-world practice. The four phases of the Quality Implementation Framework will guide implementation. Phase one focuses on identifying adaptations/strategies. Our transdisciplinary team will co-create four strategies to begin: 1) ready access to technical support, 2) scheduling flexibility, 3) broad choice of BCI activities, and 4) culturally safe care. Phase two focuses on creating a structure for implementation by formalizing plans and teams. The third phase, ongoing structure, will include monitoring and adapting strategies as needed during sequential participant enrolment. Phase four, improve future applications, will be done through evaluation outlined in outcomes below.

Home Program: Families will first complete an in-person visit to review available activities, set their first goals, and learn to use BCI independently. A BCI "kit" will be given to each family, with a headset and the equipment and software required to pursue their identified goals. Following this, families will participate in 12 virtual sessions over 3-6 months. Scheduling will be flexible to accommodate complex family needs. Daily online support will be provided via a messaging application. Participants who choose to continue using BCI beyond 12 sessions will be provided kits and supported.

Implementation Outcomes: The primary implementation outcome is the proportion of children recruited from equity-deserving groups. A baseline survey will capture comprehensive demographics. Secondary outcomes span the categories of the RE-AIM evaluation framework (Reach, Effectiveness, Adoption, Implementation, and Maintenance). These outcomes will be continuously monitored with ongoing analysis using the appropriate descriptive statistics.

Effectiveness Outcomes: The primary effectiveness outcome is achievement of child and family-identified participation-based goals, as measured by the Canadian Occupational Performance Measure (COPM). Secondary outcomes will assess quality of life, family BCI experiences (via semi-structured interviews), and health economics. Primary analyses will assess the clinical and statistical significance of pre/post changes, and secondary regression analyses will explore potential response predictors including equity-deserving factors. Inductive thematic analysis will be used for interview transcripts. Finally, brain activity via electroencephalography (EEG) data from all BCI sessions will be captured. These data will be critical to accelerate options and accuracy of pediatric-focused BCI systems.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-18 years
* Severe motor impairment including inability to walk and minimal functional hand use, and/or;
* Severe communication impairment
* Ability to follow simple instructions and attend to simple tasks
* Home environment suitable for the program based on clinician and family discussion;
* Informed assent/consent

Exclusion Criteria:

* Epileptic encephalopathy
* Unstable epilepsy, or
* Brain imaging incompatible with BCI functionality

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | Baseline and end of treatment at 6 months
  The primary effectiveness outcome is achievement of child and family-identified participation-based goals, as measured by the Canadian Occupational Performance Measure (COPM). Participants/families will set 3-5 goals, and then score the Importance, Performance, and Satisfaction with each goal on a 1-10 scale.
Implementation Reach | through study completion, an average of 2 years
  The primary implementation outcome is the proportion of children recruited from equity-deserving groups. A baseline survey will capture comprehensive demographics.

IPD SHARING:
Plan to Share IPD: Undecided